CLINICAL TRIAL: NCT06781164
Title: Examination of the Applicability and Performance of Otolaryngology Telemedicine, Telediagnostics in Establishing the Diagnosis and Therapy of Otolaryngology Diseases
Acronym: TMED_FOG_001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Collaborators: University of Szeged, Hungary (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: University of Szeged
Record Dates: First submitted 2024-12-26; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Ear Infection; Telemedicine
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- telemedicine arm (Experimental): A recording of the ear of each patient with an ear problem was taken with the device, and then they were diagnosed and prescribed therapy in the traditional way.
  Interventions: Device: telemedicine

INTERVENTIONS:
Device: telemedicine — Recording of the ear of each patient with an ear problem

SUMMARY:
System/Device name: Otoscopic recording and clinical data telemedicine software supporting its transmission and analysis.

Characteristics of the medical device:

The device is applied to an iPhone with a CE mark also from a CE-marked optical unit and the system operator, a consists of software under investigation.

DETAILED DESCRIPTION:
The detailed operation is in the user guide in Hungarian included. The device makes a video recording of the external ear canal and about the tympanic membrane, and it records clinical data (symptoms, complaints).

The telephone application sends the data through the system to a doctor, who, by analyzing them, makes a diagnosis and provides therapy.

The study is a prospective, single-arm study. The specialist treating the real patient (called doctor 2) does not see or know the diagnosis and the therapy from the telemedicine system, or the recommendation from the telemedicine The diagnosis and therapeutic treatment established by the two methods are evaluated by an independent specialist and decides whether the primary diagnosis and therapeutic treatment are the same or not in the telemedicine system.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Patients with ear complaints (especially, but not exclusively, ear pain from the ear discharge, itching, cerumen accumulation,)
* The subject communicates well with the investigator and is able to understand the requirements of the test plan and to help with compliance.

Exclusion Criteria:

* Poor general condition
* Based on the investigator's decision, a condition that directly threatens life or a symptom that corresponds to these may indicate (e.g.: Liquor dripping, massive bleeding, etc.)
* Any disease that, in the investigator's opinion, endangers the patient's health and/or contraindicates performing the test
* The examiner finds that further participation is a disadvantage for the patient for any reason;
* the patient requests the suspension of his participation orally or in writing

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the diagnoses treatments made by remote diagnostics and an on-site specialist. | 1 day
  The primary objectives of the study is: number of matching cases, measured with the similarity and matching of International Classification of Diseases (ICD) codes.
Comparison of therapy | 1 day
  Matching or similarity of prescribed therapy, e.g. same family of antibiotics , or the type of active substance. The match based on Anatomical Therapeutic Chemical (ATC) Classification

CONTACTS AND LOCATIONS:
Locations (1):
- Otorhinolaryngology and Head and Neck Surgery Clinic, Szeged, Csongrád megye, Hungary

IPD SHARING:
Plan to Share IPD: No